CLINICAL TRIAL: NCT03031002
Title: Extinction Generalization in Exposure Therapy for Spider Phobia
Brief Title: Extinction Generalization in Exposure Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Armin Zlomuzica, Dr., Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZL 59/2-2
Record Dates: First submitted 2017-01-14; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Specific Phobia
Keywords: exposure; spider phobia; generalization; extinction
MeSH Terms: conditions — Phobia, Specific; Arachnophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposure Treatment (Experimental): Participants of this arm receive two 60-minute sessions of exposure treatment for spider fear
  Interventions: Behavioral: Exposure treatment for spider fear
- No Exposure Treatment (No Intervention): Participants of this arm receive no exposure or other adequate treatment

INTERVENTIONS:
Behavioral: Exposure treatment for spider fear — Two sessions (each session = 60 minutes) of in-vivo exposure treatment (including psychoeducation) with two different spiders. Exposures comprise a hierarchy of 7 steps, to be completed with both spiders.
  Arms: Exposure Treatment

SUMMARY:
Patients with anxiety disorders oftentimes express fear responses to more than only one fear-inducing object. The principal aim of this study is to examine whether the beneficial effects of exposure on fear reduction in spider phobia can extend to stimuli which are conceptually similar to spiders (i.e. cockroaches), but have never been presented during the respective treatment.

DETAILED DESCRIPTION:
Fear extinction has evolved as the central mechanism underlying exposure-based treatments. Findings from conditioning studies indicate that fear reduction following a fear extinction procedure can generalize from the extinction stimulus to other conceptually and perceptually related stimuli. This study is aimed at translating these findings to a clinical application and will hence examine whether the basic principles of extinction generalization are applicable to exposure.

Patients with spider phobia will either receive two sessions of in-vivo exposure with spiders or no treatment. Prior to as well as after treatment, patient's fear of spiders will be assessed using the Behavioral Approach Test (BATs) and self-report questionnaires. In addition, BATs with cockroaches will be conducted to examine the effects of exposure therapy on extinction generalization.

ELIGIBILITY:
Inclusion Criteria:

* spider phobia according to Diagnostic and Statistical Manual of Mental Disorders (DSM) -IV criteria

Exclusion Criteria:

* any neurological or neuropsychiatric condition
* current behavioral or pharmacological treatment
* any mental disorder that is considered more severe than specific phobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in the Behavioral Approach Test (BAT) from pre- to posttreatment | Pre- and Posttreatment (with approximately 4 days between pre- and posttreatment)
  Behavioral Approach Tests with Spiders and Cockroaches will be conducted at pre- and posttreatment. Here, the closest proximity a participant is able to attain to the spider/cockroach will be measured.

SECONDARY OUTCOMES:
Change in Subjective Fear / Disgust during the Behavioral Approach Tests (BATs) using the Subjective Units of Distress Scale (SUDS) | Pre-and Posttreatment (with approximately 4 days between pre- and posttreatment)
  Subjective Fear / Disgust during the Behavioral Approach will be assessed at the initial and final approach distances to the spider / cockroach during the respective BATs.
Change in Heart Rate during the Behavioral Approach Tests (BATs) from pre- to posttreatment | Pre- and Posttreatment (with approximately 4 days between pre- and posttreatment)
  During each BAT with spiders and cockroaches, heart rate will be measured. In addition, a 5-minute baseline will be recorded prior to the first BAT at each assessment.
Change in the Fear of Spiders Questionnaire (FSQ) | Pre- and Posttreatment (with approximately 4 days between pre- and posttreatment)
Change in the Spider Phobia Questionnaire (SPQ) | Pre- and Posttreatment (with approximately 4 days between pre- and posttreatment)
Change in the Spider Beliefs Questionnaire (SBQ) | Pre- and Posttreatment (with approximately 4 days between pre- and posttreatment)

OTHER OUTCOMES:
Epigenetic / DNA methylation | Pre- and posttreatment (with approximately 4 days between pre- and posttreatment)
  DNA collection kits at pre- and posttreatment
Depression Anxiety Stress Scales (DASS) | Pretreatment (assessed once prior to treatment)
Questionnaire for the Assessment of Disgust Sensitivity (FEE) | Pretreatment (assessed once prior to treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Zlomuzica, Dr., Principal Investigator — Ruhr University of Bochum

IPD SHARING:
Plan to Share IPD: No